CLINICAL TRIAL: NCT06807112
Title: The Influence of Secretin Stimulated Pancreatic Secretion on Circulating Tumor DNA Expression in Patients With Pancreatic Ductal Adenocarcinoma: The Role of Biomarkers in Determining the Prognosis of Pancreatic Ductal Adenocarcinoma
Brief Title: The Influence of Secretin Stimulated Pancreatic Secretion on ctDNA Expression in Patients With Pancreatic Ductal Adenocarcinoma: The Role of Biomarkers in Determining the Prognosis of Pancreatic Ductal Adenocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital in Prague, Czech Republic (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01012025
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer
Keywords: Secretin; Panreatic ductal adenocarcinoma; Biomarker; Circulating tumor DNA
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pancreatic ductal adenocarcinoma scheduled for surgery: Both male and female patients of all age diagnosed with pancreatic ductal adenocarcinoma and indicated for surgical treatment by multidisciplinary tumor board. Patients with and without previously completed chemotherapy will be included.
  Interventions: Other: Intravenously administered secretin

INTERVENTIONS:
Other: Intravenously administered secretin — 16 micrograms of liquid secretin will be one-time intravenously administered to patients with PDAC during the first hour of surgery. Four peripheral blood samples will then be collected. Plasmatic levels of ctDNA will be measured. Plasmatic levels of biomarkers such as mRNA, miRNA, siRNA, exoRNA, S100 proteins and amino acids, isolated from the same blood samples, will be measured and analyzed in correlation to tumor volumometry, survival rate etc. in specific intervals during follow-ups.

SUMMARY:
The goal of this study is to assess the influence of pancreatic secretion stimulation by intravenously administered secretin on circulating tumor DNA in patients with pancreatic ductal adenocarcinoma. Additional aim of the study is to analyse a role of specific biomarkers in determining the prognosis of this disease. The main question o answer is:

Does intravenous secretin administration potentiate the release of circulating tumor DNA in patients with pancreatis ductal adenocarcinoma?

Additional question is:

Is there a biomarker specific and sensitive enough to help to predict the prognosis and the at the time status of the disease?

Participants scheduled for surgical treament due to pancreatic ductal adenocarcinoma will be included and stimulated with intravenously administered secretin, their peripheral blood samples will then be analyzed for ctDNA levels.

DETAILED DESCRIPTION:
Background Pancreatic ductal adenocarcinoma (PDAC) is an aggressive oncological disease with a poor prognosis and low survival rate. Due to its biological nature, it is generally challenging to accomplish early diagnostics and therefore to achieve successful therapeutic results.

Recently, many trials and studies worldwide aim at better understanding of tumor biology and providing a novel tool for diagnostics, disease monitoring and developing a targeted therapy. One of the subjects of interest happen to be the so-called liquid biopsies.

Isolation of biomarkers such as miRNA, tumor suppressor genes or amino acids from these biopsies, their analysis, quantification and incorporation into clinical oncology represents a complex issue where further research is highly required. Subjects, materials, methods A crucial prerequisite for biomarker analysis is a sufficient amount of genetic information. In our study, the effect of intravenous secretin administration on ctDNA release in patients with PDAC will be analysed. More than 90% KRAS mutation rate in patients with PDAC has been scientifically proven, therefore patients with positive KRAS mutation in their peripheral blood plasma and scheduled for surgical therapy will be included in the study.

Peripheral blood plasma of 36 patients with PDAC diagnosis will then be collected in specific intervals during the first two hours of the operation. Plasmatic levels of ctDNA in the samples will be quantified. A standardized panel of biomarkers will be designed and tested in patients with PDAC prior to surgery and in specific intervals after surgery. The results will be analyzed in correlation to minimal residual disease, survival rate and other indicators to determine the prognosis of the disease. Statistic evaluation will be done in cooperation with specialists experienced in bioinformatics and biomedical statistics.

Introduction:

Pancreatic ductal adenocarcinoma (PDAC) ranks among the most serious and aggressive malignant diseases with an unfavorable prognosis and high mortality [1,2]. Five year survival for patients with PDAC is 10 %, and ten-year survival is 6 % [3]. According to the Institute of Health Information and Statistics of the Czech Republic, incidence of PDAC in Czechia is 21.9/100000 inhabitants, prevalence is 23,2/100000 inhabitants. In addition to insufficient response to systemic chemotherapy, this statistic also contributes significantly to the difficulty of early detection of the disease due to its often asymptomatic period, while treatment methods may be significantly limited at the time of diagnosis. The indication of surgical treatment as a potentially curative method clearly depends on the established extent of the disease [4]. Currently, the worldwide monitored marker is the level of Ca19-9 in the serum, also in relation to the determination of preoperative and postoperative prognosis [5]. However, due to the lack of sufficient sensitivity and specificity for PDAC, Ca19-9 cannot be classified as a specific marker with sufficient predictive value [6]. More than three hundred markers have been proposed in various biological materials (blood, urine, feces, saliva, bile, pancreatic juice, etc.) for screening, early diagnosis, response to treatment and prognosis, but none of the biomarkers currently has a wider application in daily clinical practice [6,7].

According to recent studies, several biomarkers [6] have been identified with a high potential for further investigation in correlation with the assessment of prognosis and future use in screening in the general population [6,7,8] Early diagnosis is a key part of treatment options and the prognosis improvement in PDAC, therefore a set of biomarkers with significant potential for practical clinical use was chosen for this project to be analyzed. One of those is KRAS protooncogene from the RAS family, which is frequently mutated in PDAC [9, 10, 11, 12]. The mutated KRAS gene is about to be detected from the ctDNA isolated from the patient's plasma before and after intravenous stimulation with secretin, a hormone responsible also for pancreatic secretion [13]. We suppose that the secretin stimulation is going to potentiate the release of ctDNA.

Analysis of mutant KRAS, mRNA, miRNA, siRNA, exoRNA, S100 proteins and amino acids could therefore become an efficient hallmark in PDAC monitoring during the diagnostic - therapeutic process.

Objectives:

The aim of this project is to prove the potentiating influence of intravenous secretin stimulation on ctDNA release in patients with PDAC and thereby mediate higher plasmatic levels of ctDNA potentially usable for further analysis. Besides that, the role of KRAS mutation in ctDNA, mRNA, miRNA, siRNA, exoRNA, S100 proteins and amino acids is about to be analyzed throughout the therapeutic process to monitor the correlation of the marker levels to the standardized indicators of life expectancy, quality of life etc. at a time.

Zero hypothesis:

The plasmatic level of ctDNA after intravenous secretin administration will not be significantly higher than before the administration. The plasmatic levels of mRNA, miRNA, exogenic RNA and S100 proteins will not be significantly lower after surgery than prior to surgery and they will not show any correlation with postoperative course of the disease.

Methodology and statistic evaluation:

In the first phase, both male and female patients in any age-range diagnosed with PDAC and indicated for surgical therapy will be selected. Considering multiple blood sample collections in a short period of time, physiological effects of secretin and logistic optimization of the process, we have decided to involve the patients indicated for surgery.

Patients with tumor duplicity will be excluded. Only the patients with signed consent of participation in the study will be included. These patients' blood plasma will be collected from a peripheral vein during an outpatient visit prior to surgery and tested for the positivity of mutated KRAS gene with heteroduplex analysis using denaturing capillary electrophoresis.

36 patients with KRAS positive plasma sample will then be routinely prepared for surgery. In the first two hours of the surgical procedure, 16 micrograms of intravenous secretin will be applied. During this period of time, the intravenous secretin administration to the patient is safe and will not interfere with the surgical phase of pancreatic resection. In the interval of 3 minutes and 3x 5 minutes from the secretin application, blood samples will be collected from the peripheral vein as well by the anesthesia personnel. All blood samples will be collected to the prepared sampling kits with no need for further technical processing, transported to the laboratory and subjected for the analysis and quantification of ctDNA ant other candidate markers. In the second phase of the project, the most promising marker panels will be established based on the current knowledge and preliminary results. Blood plasma of the patients diagnosed with PDAC, indicated for surgical therapy will then be tested for the marker levels preoperatively and postoperatively before dismissal, 3, 6 and 12 months after surgery during outpatient examination. The results will then be analyzed and evaluated statistically in correlation with minimal residual disease, survival rate, quality of life and other standardized indicators to monitor the prognosis of the disease. Statistic evaluation will be realized in cooperation with specialists with a broad experience in bioinformatics and biomedical statistics.

Outcomes and significance:

Our project will provide a systematic literature review regarding liquid biopsy and biomarker analysis and its incorporation to clinical oncology in patients diagnosed with PDAC. The effect of intravenous administration of secretin on ctDNA release to patients with PDAC as an innovative method will be analyzed, potentially procuring a significantly larger amount of genetic information for biomarker analysis in these patients. Moreover, the results and outcome will help to design a panel of biomarkers and to evaluate their clinical implication in disease monitoring and prognosis evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with pancreatic ductal adenocarcinoma
* patients indicated for surgery by multidisciplinary tumor board
* patients without previously administered chemotherapy
* patients with previously administered chemotherapy

Exclusion Criteria:

* patients diagnosed with pancreatic ductal adenocarcinoma, at the time indicated for different than surgical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited as citizens of either Czech or Slovak republic, in any age-range, examined at various departments such as Gastroenterology, Surgery, Radiology in various healthcare facilities, recommended for multidisciplinary tumor board as a part of the Pancreatic Surgery Center, Department of Surgery, Military University Hospital in Prague.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2025-02-09 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Plasmatic level of circulating tumor DNA | During the surgery: 3, 8, 13, 18 minutes after secretin administration; 3, 6 and 12 months after surgery
  ng/ml

SECONDARY OUTCOMES:
Plasmatic levels of mRNA, miRNA, S100 proteins, siRNA, exoRNA. | During the surgery: 3, 8, 13, 18 minutes after secretin administration; 3, 6 and 12 months after surgery.
  ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bureš, prof., MD, CSc., FCMA, Study Director — Military University Hospital in Prague; Kristýna Pončáková, MD, Principal Investigator — Military University Hospital in Prague
Locations (1):
- Department of Surgery, Military University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sarantis P, Koustas E, Papadimitropoulou A, Papavassiliou AG, Karamouzis MV. Pancreatic ductal adenocarcinoma: Treatment hurdles, tumor microenvironment and immunotherapy. World J Gastrointest Oncol. 2020 Feb 15;12(2):173-181. doi: 10.4251/wjgo.v12.i2.173. PMID 32104548
- [Background] Ushio J, Kanno A, Ikeda E, Ando K, Nagai H, Miwata T, Kawasaki Y, Tada Y, Yokoyama K, Numao N, Tamada K, Lefor AK, Yamamoto H. Pancreatic Ductal Adenocarcinoma: Epidemiology and Risk Factors. Diagnostics (Basel). 2021 Mar 20;11(3):562. doi: 10.3390/diagnostics11030562. PMID 33804776
- [Background] Kamisawa T, Wood LD, Itoi T, Takaori K. Pancreatic cancer. Lancet. 2016 Jul 2;388(10039):73-85. doi: 10.1016/S0140-6736(16)00141-0. Epub 2016 Jan 30. PMID 26830752
- [Background] Imaoka H, Shimizu Y, Senda Y, Natsume S, Mizuno N, Hara K, Hijioka S, Hieda N, Tajika M, Tanaka T, Ishihara M, Niwa Y, Yamao K. Post-adjuvant chemotherapy CA19-9 levels predict prognosis in patients with pancreatic ductal adenocarcinoma: A retrospective cohort study. Pancreatology. 2016 Jul-Aug;16(4):658-64. doi: 10.1016/j.pan.2016.04.007. Epub 2016 Apr 22. PMID 27178104
- [Background] O'Neill RS, Stoita A. Biomarkers in the diagnosis of pancreatic cancer: Are we closer to finding the golden ticket? World J Gastroenterol. 2021 Jul 14;27(26):4045-4087. doi: 10.3748/wjg.v27.i26.4045. PMID 34326612
- [Background] Turanli B, Yildirim E, Gulfidan G, Arga KY, Sinha R. Current State of "Omics" Biomarkers in Pancreatic Cancer. J Pers Med. 2021 Feb 14;11(2):127. doi: 10.3390/jpm11020127. PMID 33672926
- [Background] Wolrab D, Jirasko R, Cifkova E, Horing M, Mei D, Chocholouskova M, Peterka O, Idkowiak J, Hrnciarova T, Kuchar L, Ahrends R, Brumarova R, Friedecky D, Vivo-Truyols G, Skrha P, Skrha J, Kucera R, Melichar B, Liebisch G, Burkhardt R, Wenk MR, Cazenave-Gassiot A, Karasek P, Novotny I, Greplova K, Hrstka R, Holcapek M. Lipidomic profiling of human serum enables detection of pancreatic cancer. Nat Commun. 2022 Jan 10;13(1):124. doi: 10.1038/s41467-021-27765-9. PMID 35013261
- [Background] Luo J. KRAS mutation in pancreatic cancer. Semin Oncol. 2021 Feb;48(1):10-18. doi: 10.1053/j.seminoncol.2021.02.003. Epub 2021 Feb 23. PMID 33676749
- [Background] Lan B, Zeng S, Grutzmann R, Pilarsky C. The Role of Exosomes in Pancreatic Cancer. Int J Mol Sci. 2019 Sep 4;20(18):4332. doi: 10.3390/ijms20184332. PMID 31487880
- [Background] Waters AM, Der CJ. KRAS: The Critical Driver and Therapeutic Target for Pancreatic Cancer. Cold Spring Harb Perspect Med. 2018 Sep 4;8(9):a031435. doi: 10.1101/cshperspect.a031435. PMID 29229669
- [Background] Afroze S, Meng F, Jensen K, McDaniel K, Rahal K, Onori P, Gaudio E, Alpini G, Glaser SS. The physiological roles of secretin and its receptor. Ann Transl Med. 2013 Oct;1(3):29. doi: 10.3978/j.issn.2305-5839.2012.12.01. PMID 25332973
- [Background] Perets R, Greenberg O, Shentzer T, Semenisty V, Epelbaum R, Bick T, Sarji S, Ben-Izhak O, Sabo E, Hershkovitz D. Mutant KRAS Circulating Tumor DNA Is an Accurate Tool for Pancreatic Cancer Monitoring. Oncologist. 2018 May;23(5):566-572. doi: 10.1634/theoncologist.2017-0467. Epub 2018 Jan 25. PMID 29371474
- See also: Citation — https://www.nature.com/articles/s41698-024-00505-0